CLINICAL TRIAL: NCT02400177
Title: Parenting Workshop on Emotion Regulation
Brief Title: Parents Workgroup About Emotion Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Antonio Hardan, Principle investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB32455
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Autism Spectrum Disorders
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Emotion regulation training (Experimental): This is a 4 sessions group workshop and 1 session individual pre-screening about parental emotion regulation and emotion co-regulation. In this study the facilitators will give information about efficient strategies to regulate parent emotions and their children's emotions.
  Interventions: Behavioral: emotion regulation training
- Control group (No Intervention): In this condition we will take all the measurement before and after the waiting list period.
  This group will go through the workshop after the measurements will be taken.

INTERVENTIONS:
Behavioral: emotion regulation training — This is a workshop for parents that help them to understand how to deal with emotions generally and specifically with their ASD children's emotion
  Other Names: Regulative Parenting
  Arms: Emotion regulation training

SUMMARY:
The purpose of this study is examine emotional regulation and reflective functioning in parents of children with Autism Spectrum Disorders (ASD) before and after an educational training (four sessions of group workshops). Our experimental aims are the following: 1) examine parental emotion regulation and reflective functioning in daily life, 2) examine child emotion regulation in their daily life 3)Learn about the training efficacy for ASD parents. This research study will help to formulate innovative treatment methods to reinforce positive emotion regulation and reflective functioning in both ASD children and their parents.

DETAILED DESCRIPTION:
The parents will answer questionnaires and Parent Development Interview (PDI) and the Five Minute Free Speech Sample (FMSS) as well as a number of other questionnaires.

Parents will be randomized between intervention group and control group. First session

* Introduction
* Setting expectations and goals
* General explanation of emotions and their development.
* How to recognize emotions? Why is it important to recognize them?
* Minding parents and child emotions. Second session
* Emotion Regulation (general explanation).
* Strategic for emotion regulation (Adults)
* Strategic for emotion regulation (children)
* Parental emotion regulation and the influence on the child emotion regulation
* Difficulties in ER among children with ASD Third session
* Three steps method: Feel, Think-Rethink, Regulate.
* Theory, explanation and implementation.
* Discussion: Role play of challenging highly affective parent-child interaction

Fourth session:

* Three steps method: Feel, Think-Rethink, Regulate.
* Theory, explanation and implementation.
* Discussion: Role play of challenging highly affective parent-child interaction The parents will do another PDI and will fill up the questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with autism ages 3-18

Exclusion Criteria:

* If they cant understand English they can not be part of the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Mentalization level | 1 month - 2 months
  By the Parent Development Interview (PDI) before and after the workshop we measure the metallization level

SECONDARY OUTCOMES:
Relationship coherence level | 1 month - 2 months
  By the FMSS (5 min speech sample)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided